CLINICAL TRIAL: NCT05294913
Title: Enhancing Emotional and Motivational Development in the University to Support Well-being and Retention in Diverse University Students
Brief Title: Enhancing Emotional and Motivational Development to Support Well-being and Retention in Diverse University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Katherine Cheng, PhD, Assistant Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2104695049
Record Dates: First submitted 2021-05-10; First posted 2022-03-24 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: emotion regulation; future-oriented motivation; salivary biomarkers; acculturative stress; salivary cortisol; C-reactive protein
MeSH Terms: conditions — Emotional Regulation | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Upon study enrollment, participants will be randomly assigned to either the placebo control group, or the intervention group. We will ask all participants to complete two waves of data collection on survey data and salivary samples (Wave 1 [W1] data collection will occur at the beginning of the semester; Wave 2 [W2] data collection will occur near the end of the semester). Between W1 and W2 data collection (circa mid-semester), each group will receive instructions on an intervention (placebo for the control group), and we will assess if there are any outcome differences between the two groups at the end of the semester.
Who Masked: Participant
Masking Description: Participants will not know which group they are assigned to. Each participant will receive a debriefing form at the end of the study for transparency, and control group participants will also receive the intervention kit at the completion of the study for equal opportunity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Contextualized Wish-Outcome-Obstacle-Plan (WOOP) intervention
- Placebo control group (Placebo Comparator)
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Contextualized Wish-Outcome-Obstacle-Plan (WOOP) intervention — This intervention will ask students to identify socio-culturally integrated academic or personal goals, so that students may be able to better strategize obstacle-overcoming to attain their future academic aspirations and modulate negative emotions or environments and associated physiological responses.
  Arms: Intervention group
Behavioral: Placebo — The placebo control group will receive a 5- to 10-minute online goal-setting video tutorial and confirm that they have completed it by filling out an online check-list.
  Arms: Placebo control group

SUMMARY:
Higher education is crucial for young adults in their intake of knowledge and skills to further their careers and reach their potentials. However, going through college is not necessarily an easy path. The purpose of this study is to enhance university students' well-being and educational experience by examining factors associated with stress and well-being.

The investigator plans to recruit eighty participants from a large public university in the US to provide survey data and saliva samples at two waves during the data collection semester (beginning and end of the semester). Survey data will include demographic information and help gauge psychosocial factors related to stress and well-being. Saliva will be tested for two biomarkers each wave of data collection, cortisol (sampling three times a day for diurnal patterns for two consecutive days) and c-reactive protein, which indicate physiological stress/immune responses. Additionally, participants be randomly assigned to an intervention (n = 40) or control group (n = 40), where the intervention group will undertake a brief intervention focused on motivation and emotion regulation circa mid-semester and the control group will receive a placebo goal-setting short training. The investigator aims to examine whether intervention efforts can enhance end-of-semester psychological and physiological well-being, and particularly, whether students from diverse backgrounds (e.g., first-generation, low-income, and/or BIPOC) can benefit from the intervention.

The investigator will use advanced quantitative data analysis (using Mplus v.8, in a structural equation modeling framework) to examine intervention efficacy and group differences. The investigator hypothesizes that those receiving the intervention will display a healthier profile at the end of the semester compared to their control group counterparts; and the investigator hypothesize students from diverse backgrounds will have significantly improved results from the intervention.

The study will allow a better understanding to crucial steps towards exploring how to improve the well-being, higher-education pipeline, and retention of students with diverse backgrounds, providing insight on how each student's university experience can be improved.

ELIGIBILITY:
Inclusion Criteria:

* participants who are currently enrolled students at a large public university in the Southwest of US.

Exclusion Criteria:

* individuals below the age of 18 or those who are not currently enrolled students at said university.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Salivary diurnal cortisol pattern change (from baseline to end-of-semester) | Salivary cortisol samples will be collected for two consecutive days per wave, three times per day (upon-awakening, 30-min after wake, and before bedtime), at Wave 1 (baseline, Week 3 of semester) and Wave 2 (end-of-semester, Week 16) of data collection
  Salivary cortisol (µg/dL) samples will be used to examine Hypothalamic-pituitary-adrenal-axis regulation and diurnal patterns of cortisol levels as a primary outcome.
Salivary C-reactive protein change (from baseline to end-of-semester) | Saliva samples will be collected for two consecutive days per wave, one time per day and averaged for reliability, at Wave 1 (baseline, Week 3 of semester) and Wave 2 (end-of-semester, circa Week 16) of data collection
  Salivary C-reactive protein (pg/mL) samples will be used to gauge participant well-being (as an inflammatory marker and risk factor for poor health)
Acculturative stress change (from baseline to end-of-semester) | Assessed once per wave at Wave 1 (baseline, circa Week 3 of semester) and Wave 2 (circa Week 16, end-of-semester) of data collection
  Acculturative stress will be assessed using the Societal, Attitudinal, Environment, and Familial Acculturation Stress scale (Mena et al., 1987), 24 items, 6-point Likert scale (0 = does not apply to 5 = extremely stressful), higher scores indicate more stress (worse outcome).
Quality of life (visual analogue) change (from baseline to end-of-semester) | Assessed once per wave at Wave 1 (baseline, circa Week 3 of semester) and Wave 2 (circa Week 16, end-of-semester) of data collection
  Quality of life will be assessed using a visual analogue (sliding scale from 0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine C Cheng, PhD, Principal Investigator — Assistant Research Professor
Locations (1):
- University of Arizona, Tucson, Arizona, United States